CLINICAL TRIAL: NCT03106597
Title: Manidipine Versus Amlodipine in Patients With Hypertension: Effects on Peripheral Edema Evaluated by Bioimpedance Analysis
Brief Title: Manidipine Versus Amlodipine in Patients With Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in enrolling subjects
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry)
Responsible Party: Principal Investigator, Eung Ju Kim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUGH15082 (MAAMA)
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
Keywords: Peripheral Edema; Bioimpedance Analysis
MeSH Terms: conditions — Hypertension | interventions — manidipine; Amlodipine

STUDY DESIGN:
Intervention Model Description: 1. Manidipine 20mg/day, Amlodipine 10mg/day
  2. Sealed envelope method randomization according to gender and age
     * 25 males under 55 years old
     * 25 males more than 55 years old
     * 25 females under 55 years old
     * 25 females more than 55 years old
Who Masked: Participant
Masking Description: Blinded-endpoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manidipine 20mg (Experimental): 50 patients will be administered orally manidipine 20mg/day after 1~2 week run-in period
  Interventions: Drug: Manidipine 20mg
- Amlodipine 10mg (Active Comparator): 50 patients will be administered orally amlodipine 10mg/day after 1~2 week run-in period
  Interventions: Drug: Amlodipine 10mg

INTERVENTIONS:
Drug: Manidipine 20mg — After a 1~2-week run-in period, patents will be randomized to receive manidipine (20 mg/day; n=50) for a 8-week open-labeled phase. Study drugs will be administered orally and once daily between 8:00am and 10:00am.
  BP, heart rate, adverse events and concomitant therapy are assessed and a physical examination is performed at each visit. A 12-lead standard ECG is obtained and hematology, clinical biochemistry and urine analysis investigations performed at the screening visit. A Bioelectrical Impedance Analysis (BIA) is undertaken at the screening visit and at the end of the 8-week treatment course. Patients have to attend the clinic visit every 4 weeks during the treatment period.
  Other Names: Madipine Tab(Manidipine Hydrochloride) 20mg (CJ)
  Arms: Manidipine 20mg
Drug: Amlodipine 10mg — After a 1~2-week run-in period, patents will be randomized to receive amlodipine (10 mg/day; n=50) for a 8-week open-labeled phase. Study drugs will be administered orally and once daily between 8:00am and 10:00am.
  BP, heart rate, adverse events and concomitant therapy are assessed and a physical examination is performed at each visit. A 12-lead standard ECG is obtained and hematology, clinical biochemistry and urine analysis investigations performed at the screening visit. A Bioelectrical Impedance Analysis (BIA) is undertaken at the screening visit and at the end of the 8-week treatment course. Patients have to attend the clinic visit every 4 weeks during the treatment period.
  Other Names: Amlodipine Pfizer 10mg (Pfizer)
  Arms: Amlodipine 10mg

SUMMARY:
The purpose of this study is to evaluate the effect of a third-generation Calcium Channel Blocker (CCB), manidipine, compared with second-generation Calcium Channel Blocker (CCB), amlodipine, on the development of peripheral edema using Direct Segmental Multi-Frequency Bioelectrical Impedance Analysis (DSM-BIA) method in patients with mild to moderate essential hypertension. Investigator expects this study could show more objective evidence of better safety of manidipine compared with amlodipine for peripheral edema.

DETAILED DESCRIPTION:
Dihydropyridine Calcium Channel Blockers (CCBs) are one of the most commonly used potent antihypertensive agents. Their vasodilatory effects are associated with Adverse Effects (AEs) such as peripheral edema, headache and flushing.

The incidence of peripheral edema with Calcium Channel Blocker (CCB) is 6% in a recent systematic review and is clearly dose-dependent and more common in women, in obese and in elderly hypertensives. Peripheral edema could be a cause for poor persistence with therapy or antihypertensive treatment withdrawal and has a deleterious impact on health-related quality of life.

A recent meta-analysis of head-to-head trials to compare the efficacy and safety profile of manidipine and amlodipine showed significantly better safety of manidipine: the Relative Risk (RR) for adverse event was 0.69 (0.56-0.85), and particularly for ankle edema Relative Risk (RR) was 0.35 (0.22-0.54).

Although peripheral edema is an important issue in Calcium Channel Blocker (CCB) treatment, techniques (e.g, ankle-foot volume using a water displacement measurement, plethysmography, and pretibial subcutaneous tissue pressure) for the objective measurement are not generally available in a clinical setting. Most clinical studies relied on self-report of peripheral edema that is not a reliable objective method.

Recently, Bioelectrical Impedance Analysis (BIA) has become increasingly popular for estimating body composition, including Extracellular Water (ECW) and Intracellular Water (ICW), fat mass and fat-free mass. Mechanistically, the Calcium Channel Blocker (CCB)-related peripheral edema is likely due to distal arteriolar dilatation with capillary leak to tissue spaces. Because BIA method can measure the edema as the ratio of Extracellular Water (ECW) to Total Body Water (TBW), it may reflect the Calcium Channel Blocker (CCB)-related edema. Moreover, the Direct Segmental Multi-frequency Bioelectrical Impedance Analysis (DSM-BIA) has been validated to assess segmental body (i.e., trunk, arms and legs) composition in addition to total body composition and can provide segmental edema score as well as total edema score. This new, previously not reported method is expected to provide more objective and precise data for peripheral edema.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of 20 and 80 years with uncomplicated essential hypertension are eligible.
* Inclusion criteria requires that patients have either stage I or stage II hypertension (mean sitting systolic Blood Pressure (BP) 140-179 mmHg, diastolic BP 90-109 mmHg).
* The patients are newly diagnosed or known hypertensive subjects who were not taking antihypertensive agents for more than the last 4 weeks.

Exclusion Criteria:

* Patients are excluded from the study if they have any evidence of clinically significant concurrent medical conditions including cardiac, renal, hepatic, gastrointestinal, or endocrinologic disease.
* Patients are also excluded if they have known hypersensitivity or serious drug reactions to Calcium Channel Blockers (CCBs), any evidence of prior deep vein thrombosis, lymphatic disease, or concurrent requirement for medications that could affect Blood Pressure (BP) or salt and water retention (e.g, nonsteroidal antinflammatory drugs, estrogen containing drugs).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Change in leg edema score (Extracellular Water(ECW) to Total Body Water(TBW)) | Up to 8 weeks

SECONDARY OUTCOMES:
Changes in segmental (each arm/leg, trunk) edema score | Up to 8 weeks
Changes in Blood Pressure (BP) | Up to 8 weeks
Incidences of AEs | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eung Ju Kim, MD, Principal Investigator — Professor
Locations (3):
- South Korea (3):
  - Yonsei University Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Wonju Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richy FF, Laurent S. Efficacy and safety profiles of manidipine compared with amlodipine: a meta-analysis of head-to-head trials. Blood Press. 2011 Feb;20(1):54-9. doi: 10.3109/08037051.2010.518670. Epub 2010 Oct 14. PMID 20945994
- [Background] Opie LH. Calcium channel antagonists. Part IV: Side effects and contraindications drug interactions and combinations. Cardiovasc Drugs Ther. 1988 Jul;2(2):177-89. doi: 10.1007/BF00051233. PMID 3154704
- [Background] Makani H, Bangalore S, Romero J, Wever-Pinzon O, Messerli FH. Effect of renin-angiotensin system blockade on calcium channel blocker-associated peripheral edema. Am J Med. 2011 Feb;124(2):128-35. doi: 10.1016/j.amjmed.2010.08.007. PMID 21295192
- [Background] Messerli FH, Oparil S, Feng Z. Comparison of efficacy and side effects of combination therapy of angiotensin-converting enzyme inhibitor (benazepril) with calcium antagonist (either nifedipine or amlodipine) versus high-dose calcium antagonist monotherapy for systemic hypertension. Am J Cardiol. 2000 Dec 1;86(11):1182-7. doi: 10.1016/s0002-9149(00)01199-1. PMID 11090788
- [Background] Fogari R. Ankle oedema and sympathetic activation. Drugs. 2005;65 Suppl 2:21-7. doi: 10.2165/00003495-200565002-00004. PMID 16398059
- [Background] Weir MR, Rosenberger C, Fink JC. Pilot study to evaluate a water displacement technique to compare effects of diuretics and ACE inhibitors to alleviate lower extremity edema due to dihydropyridine calcium antagonists. Am J Hypertens. 2001 Sep;14(9 Pt 1):963-8. doi: 10.1016/s0895-7061(01)02167-7. PMID 11587165
- [Background] Fogari R, Malamani G, Zoppi A, Mugellini A, Rinaldi A, Fogari E, Perrone T. Effect on the development of ankle edema of adding delapril to manidipine in patients with mild to moderate essential hypertension: a three-way crossover study. Clin Ther. 2007 Mar;29(3):413-8. doi: 10.1016/s0149-2918(07)80079-8. PMID 17577462
- [Background] Seo HS, Kim EJ, Kim SW, Im SI, Na JO, Choi CU, Lim HE, Won Kim J, Rha SW, Park CG. Extracellular fluid adjusted for body size is contracted in hypertension. Hypertens Res. 2013 Oct;36(10):916-21. doi: 10.1038/hr.2013.68. Epub 2013 Jul 11. PMID 23842617
- [Background] Ling CH, de Craen AJ, Slagboom PE, Gunn DA, Stokkel MP, Westendorp RG, Maier AB. Accuracy of direct segmental multi-frequency bioimpedance analysis in the assessment of total body and segmental body composition in middle-aged adult population. Clin Nutr. 2011 Oct;30(5):610-5. doi: 10.1016/j.clnu.2011.04.001. Epub 2011 May 8. PMID 21555168
- [Background] Schoeller DA, Alon A, Manekas D, Mixson LA, Lasseter KC, Noonan GP, Bolognese JA, Heymsfield SB, Beals CR, Nunes I. Segmental bioimpedance for measuring amlodipine-induced pedal edema: a placebo-controlled study. Clin Ther. 2012 Mar;34(3):580-92. doi: 10.1016/j.clinthera.2012.01.018. Epub 2012 Mar 3. PMID 22385927